CLINICAL TRIAL: NCT02038959
Title: Using Technology to Deliver Multi-disciplinary Care to Individuals With Parkinson Disease in Their Homes: the Connect.Parkinson Study
Brief Title: Connect.Parkinson: Connecting Individuals With Parkinson Disease to Specialists in Their Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Parkinson Foundation (Other)
Responsible Party: Principal Investigator, Ray Dorsey, Director, Center for Human Experimental Therapeutics; Professor of Neurology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AD-12-11-4701
Record Dates: First submitted 2014-01-08; First posted 2014-01-17 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Parkinson's; Parkinson's disease; telemedicine; virtual visits; video calls; video conferencing; virtual house calls
MeSH Terms: conditions — Parkinson Disease | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care and Educational Materials (No Intervention): Participants with Parkinson disease will receive educational materials from the National Parkinson Foundation, complete a baseline assessment survey and virtual visit with a physician independent rater, then continue with their usual care in their communities for the duration of the study. After 12 months, they will have another virtual study assessment with an independent rater, after which they will receive a free, one-time virtual consultation with a Parkinson disease specialist in their state.
- Virtual Visits and Educational Materials (Experimental): Participants with Parkinson disease randomized to the virtual visit intervention will receive educational materials from the National Parkinson Foundation, complete a baseline assessment and virtual study assessment with a physician independent rater, and then receive four virtual care visits with a Parkinson disease specialist in their state. Specialists will provide recommendations for care to participants and their designated local health care provider. At 12 months, these individuals will again be assessed by the independent rater, who will be blind to treatment assignment.
  Interventions: Other: Virtual Visits

INTERVENTIONS:
Other: Virtual Visits — Virtual visits will be completed using HIPAA-compliant video conferencing software from SBR Health and Vidyo, designed specifically for use in the healthcare industry. The software is available for Windows and Mac OS, as well as iOS devices (iPad and iPhone).
  Other Names: Telemedicine; Teleneurology; Video call; Video conferencing
  Arms: Virtual Visits and Educational Materials

SUMMARY:
Connect.Parkinson is a randomized comparative effectiveness study, comparing usual care enhanced with educational materials to usual care, educational materials, and the delivery of specialty care via telemedicine into patient's homes. The study's specific aims are the following:

1. To demonstrate the feasibility of using telemedicine to deliver specialty care into the homes of individuals with Parkinson disease who have limited access to care;
2. To show that such an approach can improve quality of life;
3. To establish that the telemedicine can enhance the quality of care; and
4. To demonstrate that this remote approach to care saves time, reduces travel, and decreases care partner burden.

DETAILED DESCRIPTION:
Connect.Parkinson is a national study examining the feasibility and effectiveness of using video calls to bring expert Parkinson disease care directly into patients' homes. Currently, access to care for Parkinson disease is limited by distance, disability, and the distribution of doctors. Approximately 200 individuals with Parkinson disease (who due to distance, disability, disparity, or doctor distribution have limited access to care) will be randomized to one of two arms in this comparative effectiveness study. The first (control) arm will be the individual's "usual care" supplemented by educational materials on their condition. This usual care may include care from a generalist, care from a neurologist, or in-person care from a Parkinson specialist. The care received by the control group will vary but will be an accurate reflection of usual care in this country. The second (intervention) arm will be usual care supplemented by educational materials and care from a Parkinson disease specialist delivered via web-based video conferencing into the patient's home. The participants will also be asked with they have a primary care partner, and care partners will be invited to enroll, for a total of approximately 400 participants.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinically diagnosed Idiopathic Parkinson disease in the judgment of the independent rater
* No better alternative explanation for the parkinsonism
* Access to a non-public, internet-enabled device (e.g., computer, tablet computer, smart phone) that has the capacity for web-based video conferencing
* Be physically located at time visits are conducted in a state where the participating physician is licensed to practice medicine
* Have a local care provider that the study team can contact
* Live at home, in a senior housing complex, or assisted living facility
* Be fluent in English (all participating states) or Spanish (participants in Florida and Massachusetts only)
* Willing and able to provide informed consent
* Care partner (if applicable) must be able and willing to provide informed consent to participate if he or she so chooses.

Exclusion Criteria:

* Currently hospitalized
* Condition (e.g., prominent psychosis) that precludes study participation as identified by the medical professional (site investigator or nurse).
* Participation in another telemedicine study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Ray Dorsey, MD, MBA, Principal Investigator — University of Rochester
Locations (20):
- United States (20):
  - University of California San Francisco, San Francisco, California
  - The Parkinson's Institute and Clinical Center, Sunnyvale, California
  - University of Florida, Gainsville, Florida
  - University of Miami, Miami, Florida
  - Georgia Regents University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Struthers Parkinson Center, Golden Valley, Minnesota
  - The Mayo Clinic, Rochester, Minnesota
  - Northshore Long Island Jewish - Feinstein Institute, Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Northwest Neurological, PLLC, Spokane, Washington

REFERENCES:
- [Background] Dorsey ER, Venkataraman V, Grana MJ, Bull MT, George BP, Boyd CM, Beck CA, Rajan B, Seidmann A, Biglan KM. Randomized controlled clinical trial of "virtual house calls" for Parkinson disease. JAMA Neurol. 2013 May;70(5):565-70. doi: 10.1001/jamaneurol.2013.123. PMID 23479138
- [Background] Grana MJ, Bull MT, Venkataraman V, Dorsey ER, Biglan KM. Web-based clinical assessments for Parkinson's disease: reliable and feasible. Mov Disord. 2012 Sep 15;27(11):1466. doi: 10.1002/mds.25121. Epub 2012 Sep 18. No abstract available. PMID 22991090
- [Background] Abdolahi A, Scoglio N, Killoran A, Dorsey ER, Biglan KM. Potential reliability and validity of a modified version of the Unified Parkinson's Disease Rating Scale that could be administered remotely. Parkinsonism Relat Disord. 2013 Feb;19(2):218-21. doi: 10.1016/j.parkreldis.2012.10.008. Epub 2012 Oct 25. PMID 23102808
- [Background] Willis AW, Schootman M, Tran R, Kung N, Evanoff BA, Perlmutter JS, Racette BA. Neurologist-associated reduction in PD-related hospitalizations and health care expenditures. Neurology. 2012 Oct 23;79(17):1774-80. doi: 10.1212/WNL.0b013e3182703f92. Epub 2012 Oct 10. PMID 23054239
- [Background] Willis AW, Schootman M, Evanoff BA, Perlmutter JS, Racette BA. Neurologist care in Parkinson disease: a utilization, outcomes, and survival study. Neurology. 2011 Aug 30;77(9):851-7. doi: 10.1212/WNL.0b013e31822c9123. Epub 2011 Aug 10. PMID 21832214
- [Background] Venkataraman V, Donohue SJ, Biglan KM, Wicks P, Dorsey ER. Virtual visits for Parkinson disease: A case series. Neurol Clin Pract. 2014 Apr;4(2):146-152. doi: 10.1212/01.CPJ.0000437937.63347.5a. PMID 24790799
- [Background] Achey MA, Beck CA, Beran DB, Boyd CM, Schmidt PN, Willis AW, Riggare SS, Simone RB, Biglan KM, Dorsey ER. Virtual house calls for Parkinson disease (Connect.Parkinson): study protocol for a randomized, controlled trial. Trials. 2014 Nov 27;15:465. doi: 10.1186/1745-6215-15-465. PMID 25431346
- [Background] Achey MA, Beck CA, Beran DB, Boyd CM, Schmidt PN, Willis AW, Riggare SS, Simone RB, Biglan KM, Dorsey ER. Erratum To: Virtual house calls for Parkinson disease (Connect.Parkinson): study protocol for a randomized, controlled trial. Trials. 2016 Jan 5;17:7. doi: 10.1186/s13063-015-0984-7. No abstract available. PMID 26733455
- [Background] Dorsey ER, Achey MA, Beck CA, Beran DB, Biglan KM, Boyd CM, Schmidt PN, Simone R, Willis AW, Galifianakis NB, Katz M, Tanner CM, Dodenhoff K, Ziman N, Aldred J, Carter J, Jimenez-Shahed J, Hunter C, Spindler M, Mari Z, Morgan JC, McLane D, Hickey P, Gauger L, Richard IH, Bull MT, Mejia NI, Bwala G, Nance M, Shih L, Anderson L, Singer C, Zadikoff C, Okon N, Feigin A, Ayan J, Vaughan C, Pahwa R, Cooper J, Webb S, Dhall R, Hassan A, Weis D, DeMello S, Riggare SS, Wicks P, Smith J, Keenan HT, Korn R, Schwarz H, Sharma S, Stevenson EA, Zhu W. National Randomized Controlled Trial of Virtual House Calls for People with Parkinson's Disease: Interest and Barriers. Telemed J E Health. 2016 Jul;22(7):590-8. doi: 10.1089/tmj.2015.0191. Epub 2016 Feb 17. PMID 26886406
- [Background] Daschle T, Dorsey ER. The return of the house call. Ann Intern Med. 2015 Apr 21;162(8):587-8. doi: 10.7326/M14-2769. No abstract available. PMID 25894028
- [Background] Dorsey ER, Topol EJ. State of Telehealth. N Engl J Med. 2016 Jul 14;375(2):154-61. doi: 10.1056/NEJMra1601705. No abstract available. PMID 27410924
- [Derived] Beck CA, Beran DB, Biglan KM, Boyd CM, Dorsey ER, Schmidt PN, Simone R, Willis AW, Galifianakis NB, Katz M, Tanner CM, Dodenhoff K, Aldred J, Carter J, Fraser A, Jimenez-Shahed J, Hunter C, Spindler M, Reichwein S, Mari Z, Dunlop B, Morgan JC, McLane D, Hickey P, Gauger L, Richard IH, Mejia NI, Bwala G, Nance M, Shih LC, Singer C, Vargas-Parra S, Zadikoff C, Okon N, Feigin A, Ayan J, Vaughan C, Pahwa R, Dhall R, Hassan A, DeMello S, Riggare SS, Wicks P, Achey MA, Elson MJ, Goldenthal S, Keenan HT, Korn R, Schwarz H, Sharma S, Stevenson EA, Zhu W; Connect.Parkinson Investigators. National randomized controlled trial of virtual house calls for Parkinson disease. Neurology. 2017 Sep 12;89(11):1152-1161. doi: 10.1212/WNL.0000000000004357. Epub 2017 Aug 16. PMID 28814455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with Parkinson disease were recruited and enrolled remotely and sent educational materials about Parkinson disease created by the National Parkinson Foundation. Recruitment for the study began in February 2014.
Pre-assignment Details: 272 individuals were referred to 18 sites to be consented. Two hundred ten individuals with Parkinson disease enrolled in the study, and 195 were eventually randomized.
Period: Overall Study
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Started | 98 | 97
Completed | 92 | 89
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials | Total
Number analyzed (Participants) | 98 | 97 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.5) | 65.9 (7.8) | 66.4 (8.1)
Gender [Count of Participants; unit: Participants]
  Female | 42 | 49 | 91
  Male | 56 | 48 | 104
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 97 | 195
Minutes spent with Parkinson disease provider [Median (Inter-Quartile Range); unit: minutes] — Time spent with the provider at the participants last appointment was collected in minutes. At baseline this would be the time the participant spent with their provider at their last appointment prior to enrolling in the study.
  minutes | 30 [20 to 45] | 30 [20 to 45] | 30 [20 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Virtual Visits for Parkinson Disease
Description: Feasibility of virtual visits will be determined by the number of participants who complete at least one virtual visit successfully.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 98 | 97
participants | 0 | 95

2. Primary Outcome: Change From Baseline in the Quality of Life Measured by Parkinson Disease Questionnaire 39
Description: Assessed as the change in quality of life, measured by the Parkinson Disease Questionnaire 39 (PDQ-39). The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month. Assesses how often patients experience difficulties across the 8 quality of life dimensions. Assesses impact of Parkinson's Disease (PD) on specific dimensions of functioning and well-being. The score ranges from 0-100 with lower scores reflecting better quality of life.
Time Frame: Baseline to One year
Population: Data was not collected on 17 participants in the usual care arm and 18 participants in the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 81 | 79
units on a scale | -0.7512 (0.9472) | -0.4123 (1.0029)
Statistical Analysis 1: Comparison: Usual Care and Educational Materials vs Virtual Visits and Educational Materials; Test type: Superiority or Other; p > 0.05, ANCOVA

3. Secondary Outcome: Change in EQ-5D Index Value
Description: EuroQol five dimensions questionnaire (EQ-5D) is a standardized instrument for measuring generic health status. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale ranges from 11111 to 55555 with higher numbers indicating worse health status. The five-digit descriptors are converted to EQ-5D Index Values, which range from -0.109 (corresponding to 55555, the worst possible health) to 1.000 (corresponding to 11111, the best possible health).
Time Frame: baseline to one year
Population: Data was not collected in 6 participants from the usual care arm and 9 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 92 | 88
units on a scale | -0.04122 (0.01074) | -0.02728 (0.01139)

4. Secondary Outcome: Change in Montreal Cognition Assessment
Description: We will assess changes in cognition from baseline to the end of the study using the Montreal Cognitive Assessment (MoCA), administered remotely. The scale ranges from 0-30 with higher numbers indicating better cognition.
Time Frame: baseline to one year
Population: Data was not collected on 6 participants in the usual care arm and 9 participants in the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 92 | 88
units on a scale | 0.2072 (0.243) | 0.6485 (0.2566)

5. Secondary Outcome: Change in Parkinson Disease Rating Scale (MDS-UPDRS) Part IA
Description: Parkinson disease clinical characteristics will be assessed by a physician independent rater, blinded to treatment group, at baseline and at the conclusion of the study, using the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS). Part I concerns nonmotor experiences of daily living. The scale ranges from 0 to 24 with higher numbers indicated more severe disease.
Time Frame: baseline to one year
Population: Data was not collected in 6 participants from the usual care arm and 8 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 92 | 89
units on a scale | -1.0122 (0.2979) | -0.8546 (0.3117)

6. Secondary Outcome: Change in Patient Assessment of Chronic Illness Care
Description: We will assess change in the perceived quality of care using the Patient Assessment of Chronic Illness Care (PACIC). Each scale is scored by averaging the items completed within that scale, and the overall PACIC is scored by averaging scores across all 20 items. The scale ranges from 1-5 with higher scores indicating better care by the health team.
Time Frame: baseline to one year
Population: Data was not collected in 16 participants from the usual care arm and 12 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 82 | 85
units on a scale | 0.2456 (0.1001) | 0.2795 (0.1035)

7. Secondary Outcome: Minutes Spend on Last Parkinson's Disease Provider Visit
Time Frame: One year
Population: Data was not collected on 10 participants in the usual care arm and 28 participants in the virtual visits arm.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 88 | 69
minutes | 30 [20 to 45] | 30 [20 to 40]
Statistical Analysis 1: Comparison: Usual Care and Educational Materials vs Virtual Visits and Educational Materials; Test type: Superiority or Other; p < 0.0001, ANCOVA

8. Secondary Outcome: Change in Parkinson Disease Rating Scale (MDS-UPDRS) Part IB
Description: Parkinson disease clinical characteristics will be assessed by a physician independent rater, blinded to treatment group, at baseline and at the conclusion of the study, using the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS). Part I concerns nonmotor experiences of daily living. The scale ranges from 0 to 52 with higher numbers indicated more severe disease.
Time Frame: baseline to one year
Population: Data was not collected in 11 participants from the usual care arm and 7 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 87 | 90
units on a scale | 0.389 (0.3701) | 0.1243 (0.3786)

9. Secondary Outcome: Change in Parkinson Disease Rating Scale (MDS-UPDRS) Part 2
Description: Parkinson disease clinical characteristics will be assessed by a physician independent rater, blinded to treatment group, at baseline and at the conclusion of the study, using the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS). Part II concerns motor experiences of daily living. The scale ranges from 0 to 52 with higher numbers indicated more severe disease.
Time Frame: baseline to one year
Population: Data was not collected in 12 participants from the usual care arm and 7 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 86 | 90
units on a scale | -0.3266 (0.5084) | 0.1378 (0.512)

10. Secondary Outcome: Change in Parkinson Disease Rating Scale (MDS-UPDRS) Part 3
Description: Parkinson disease clinical characteristics will be assessed by a physician independent rater, blinded to treatment group, at baseline and at the conclusion of the study, using the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS). Part III is retained as the motor examination. The scale ranges from 0 to 108 with higher numbers indicated more severe disease.
Time Frame: baseline to one year
Population: Data was not collected in 9 participants from the usual care arm and 9 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 89 | 88
units on a scale | -4.9164 (0.9782) | -5.7495 (1.0106)

11. Secondary Outcome: Change in Parkinson Disease Rating Scale (MDS-UPDRS) Part 4
Description: Parkinson disease clinical characteristics will be assessed by a physician independent rater, blinded to treatment group, at baseline and at the conclusion of the study, using the Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS). Part IV concerns motor complications. The scale ranges from 0 to 24 with higher numbers indicated more severe disease.
Time Frame: baseline to one year
Population: Data was not collected in 6 participants from the usual care arm and 9 participants from the virtual visits arm.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Number analyzed (Participants) | 92 | 88
units on a scale | -0.2075 (0.4042) | -0.1825 (0.425)

ADVERSE EVENTS:
Arm/Group | Usual Care and Educational Materials | Virtual Visits and Educational Materials
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/97
Other Adverse Events (participants affected / at risk) | 0/98 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes